CLINICAL TRIAL: NCT05401825
Title: Antenatal COVID 19 VACCINATION and Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: 2311
Record Dates: First submitted 2022-06-01; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Effect of Drug

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: pfizer, astrazeneca,moderna,sinofac — effect of COVID 19 vaccination on pregnancy outcomes

SUMMARY:
Effect of COVID 19 vaccinations on pregnancy outcomes must be clear and identified to detect their safty

DETAILED DESCRIPTION:
in this study we will discuss side effects of COVID 19 vaccine on pregnant women including the incidence of miscarrage , intrauterine fetal deaths, liquor abnormalities, preeclampsia, accidental hemorrhage , we also will follow up pregnant women who received any type of COVID 19 vaccine till delivery and discuss the effect of the vaccine on fetus and newborn

ELIGIBILITY:
Inclusion Criteria:

* pregnant women aged 18 years or older who received any type of COVID 19 vaccine during current pregnancy

Exclusion Criteria:

* comorbidities,women who refused participqtion,pregnant women with previous COVID 19 infection during current pregnancy

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant ladies received COVID 19 vaccine during pregnancy
Study Population: pregnant women aged 18 years or older who received any type of COVID 19 vaccine during current pregnancy
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
pregnancy loss | in first, second, third trimester
  miscarrage or intrauterine fetal death

SECONDARY OUTCOMES:
fetal malformations | at each trimester
  detected by detailed anomaly scan
pregnancy related hypertensive disorders | starting from 20 weeks of gestation
  blood pressure higher than 140/90mmHg starting from 20 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mamdouh, assistant professor, Study Director — Ainshams university; Walid H Eltantawy, professor, Study Director — Ainshams university
Locations (1):
- Ainshams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided